CLINICAL TRIAL: NCT05821660
Title: Metabolic Effects of a Five-day Remotely Delivered Hypocaloric and Ketogenic Program in Healthy Subjects
Brief Title: Fastreset Study: Metabolic Effects of a Five-day Remotely Delivered Hypocaloric and Ketogenic Program
Acronym: Fastreset
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buchinger Wilhelmi Development & Holding GmbH (Other)
Collaborators: Buchinger Wilhelmi Clinic (Unknown); King's College London (Other); MVZ Labor Ravensburg GbR (Unknown); Synlab Málaga (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F-2023-014
Record Dates: First submitted 2023-03-22; First posted 2023-04-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy Nutrition; Healthy Lifestyle
Keywords: hypocaloric and ketogenic diet; intestinal microbiota; inflammatory status

STUDY DESIGN:
Intervention Model Description: Prospective, two-arm interventional study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Five-day hypocaloric and ketogenic programme (Experimental): The group will receive a five-day remotely delivered hypocaloric and ketogenic programme followed by a four-day food reintroduction period
  Interventions: Other: Five-day hypocaloric and ketogenic programme
- Control (No Intervention): The group will maintain their habitual diet

INTERVENTIONS:
Other: Five-day hypocaloric and ketogenic programme — Dietary intervention
  Other Names: Buchinger Wilhelmi Fastingbox
  Arms: Five-day hypocaloric and ketogenic programme

SUMMARY:
The aim of this study is to assess changes in body and metabolism caused by this new five-day hypocaloric and ketogenic programme

DETAILED DESCRIPTION:
Therapeutic effects of fasting are increasingly documented. Recent studies on a cohort of subjects doing a long-term fasting lasting from 4 days to several weeks demonstrated beneficial effects on health and well-being. In recent studies on the therapeutic efficacy of the Buchinger Wilhelmi fasting program, long-term fasting significantly improved risk factors for a variety of chronic diseases including hypertension even in medicated subjects, liver steatosis, inflammation, oxidative stress and lipoprotein distribution.

There is an increasing demand for dietary interventions which can be delivered at home. This has been amplified by the Coronavirus-19 disease (COVID-19) pandemic during which many countries kept their population in lockdown at home in isolation. The COVID-19 pandemic has also influenced the lifestyle of individuals, with an increased consumption of unhealthy food and a sedentary behaviour resulting in mental (anxiety, depression, and others) and physical (weight gain, rise in blood pressure) health issues. In order to adapt to this new context, the Buchinger Wilhelmi Clinics have created a hypocaloric, ketogenic program with interval fasting.

The five-day programme is designed to be easily integrated into everyday life and can be applied several times a year. The programme is based on ready-to-eat soups made with locally sourced organic ingredients. The ingredients represent a total daily intake of around 600 kcal per day - with a high share of fats and a limited quantity of carbohydrates and proteins. Minerals and micronutrients used at the Buchinger Wilhelmi Clinics are also supplied. Although the comprehensive medical care and assistance offered at the clinics cannot be replicated, medical professionals are available to support the customers remotely.

The investigators hypothesise that the metabolic changes caused by this new five-day programme can be similar to a short-term fast. In order to test this hypothesis, the investigators will perform a two-arm randomized controlled trial in which a group of participants will perform the five-day Fastingbox programme and a group of participants will receive an eucaloric diet as a control group.

ELIGIBILITY:
Exclusion Criteria:

* Not able to sign the informed consent
* diagnosticated with cachexia, anorexia, nervosa, advanced kidney, liver or cerebrovascular insufficiency.
* Intake of antibiotics up to 2 months prior the study
* Medicated high blood pressure
* Diagnosed hyperuricemia
* Diagnosed diabetes mellitus type I and II
* Diagnosed kidney stone
* Active malignant diseases
* Known substance addiction
* Pregnancy or breastfeeding
* Participation in another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | through study completion (11 subsequent days as well as one month afterwards)
  in kg
Changes in systolic blood pressure | through study completion (11 subsequent days as well as one month afterwards)
  in mmHg
Changes in diastolic blood pressure | through study completion (11 subsequent days as well as one month afterwards)
  in mmHg

SECONDARY OUTCOMES:
Changes in acetoacetic acid | through study completion (11 subsequent days as well as one month afterwards)
  measured by nitroprussid test in urine in mg/dL
Changes in total cholesterol | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (photometry)
Changes in HDL-C | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (elimination/catalase)
Changes in LDL-C | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (elimination/catalase)
Changes in triglycerides | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (GPO, trinder without serum blank) in mmol/l
Changes in glucose | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (hexokinase) in mmol/l
Changes in HbA1c | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (HPLC) in %
Changes in Insulin | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (CLIA) in mU/l
Changes in total antioxidant capacity | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique
Changes in lipidperoxidation | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (in µmol/l)
Changes in well-being | through study completion (11 subsequent days as well as one month afterwards)
  WHO-5 well-being index
Changes in ESR | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in mm/h by kinetic flow analysis in capillaries on a photometric basis
Changes in CRP | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique
Changes in IL-6 | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (ECLIA)
Changes in IL-10 | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique
Changes in TNF-a | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (CLIA)
Changes in gut microbiome composition | At baseline, first stool after 9 days as well as 1 month afterwards
  Shotgun metagenomics, qPCR, SCFA

OTHER OUTCOMES:
Changes in body mass index | through study completion (11 subsequent days as well as one month afterwards)
  in kg/m²
Changes in abdominal circumference | through study completion (11 subsequent days as well as one month afterwards)
  in cm
Changes in resting heart frequency | through study completion (11 subsequent days as well as one month afterwards)
  in beats/min
Changes in leucocytes | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (electronic count)
Changes in erythrocytes | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (electronic count)
Changes in haemoglobin | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (photometry)
Changes in haematocrit | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (electronic count)
Changes in MCV | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (ELISA)
Changes in MCH | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique
Changes in MCHC | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique
Changes in thrombocytes | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (electronic count)
Changes in INR | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (coagulometry) in sec
Changes in PTT | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (coagulometry) in sec
Changes in kidney parameters | At baseline, after 5 and 9 days as well as 1 month afterwards
  blood parameters: uric acid, urea, creatinine in mg/dl
Changes in uric acid | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (enzymatic/uricase/peroxidas) in mg/dl
Changes in urea | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (GLDH) in mg/dl
Changes in creatinine | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (creatininase) in mg/dl
Changes in GOT | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (IFCC method) in U/l
Changes in GPT | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (IFCC method) in U/l
Changes in GGT | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (IFCC modified) in U/l
Changes in AP | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique in U/l
Changes in sodium | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (potentiometric, ISE) in mmol/l
Changes in potassium | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (potentiometric, ISE) in mmol/l
Changes in calcium | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (CPC) in mmol/l
Changes in magnesium | At baseline, after 5 and 9 days as well as 1 month afterwards
  measured in serum by a routine technique (ICPMS) in mmol/l
Changes in continous glucose monitoring | At baseline, after 5 and 9 days as well as 1 month afterwards
  glucose level in mg/dl
Changes in physical activity level | At baseline, after 5 and 9 days as well as 1 month afterwards
  questionnaires: International Physical Activity Questionnaire (IPAQ) 150min./week of exercise is considered sufficient physical activity
Changes in sleep quality | At baseline, after 5 and 9 days as well as 1 month afterwards
  questionnaires: Pittsburgh Sleep Quality Index (PSQI), score ranging from 0 to 21, where lower scores denote a healthier sleep quality
Changes in processed food consumption | At baseline, after 5 and 9 days as well as 1 month afterwards
  questionnaire: highly processed food consumption (sQ-HPF)
Changes in physical well-being | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in emotional well-being | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in energy level | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in cravings | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in feeling bloated | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in feeling cold | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in tiredness | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in muscle weakness | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in back pain | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in headache | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in hunger | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in anxiety | through study completion (11 subsequent days as well as one month afterwards9
  measured by visual scale (0-10)
Changes in digestive problems | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10)
Changes in optimism | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-4)
Changes in relaxation | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-4)
Changes in clear thinking | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-4)
Changes in confidence | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-4)
Changes in happiness | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-4)
Changes in physical activity | through study completion (11 subsequent days as well as one month afterwards)
  measured by visual scale (0-10) and absolut numbers
Ethnicity | baseline
  Caucasian, Hispanic, African American, Asian, others
Smoking | baseline
  status: never, former, current, flatmate
Alcohol consumption | baseline, after 5 and 9 days as well as 1 month afterwards
  number of glasses: wine, beer, spirits
Changes in stress level | baseline, after 5 and 9 days as well as 1 month afterwards
  measured by visual scale (0-10)
Changes in energy level | baseline, after 5 and 9 days as well as 1 month afterwards
  measured by visual scale (0-10)
Changes in pain level | baseline, after 5 and 9 days as well as 1 month afterwards
  measured by visual scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Wilhelmi de Toledo, Dr., Principal Investigator — Buchinger Wilhelmi
Locations (1):
- Buchinger Wilhelmi Clinic, Überlingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided